CLINICAL TRIAL: NCT05280535
Title: Dual Use of ENDS and Combustible Cigarettes: Shared, Distinct, and Cross-Conditioned Processes
Brief Title: Dual Use of ENDS and Combustible Cigarettes
Acronym: DUET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alexander Sokolovsky, Assistant Professor, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2003002659; 1K08DA048137-01A1 (NIH)
Record Dates: First submitted 2022-01-25; First posted 2022-03-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Smoking, Cigarette; Electronic Cigarette Use
Keywords: cigarette; e-cigarette; ENDS; electronic nicotine delivery system; smoking; vaping; attentional bias; cue reactivity; negative affect; craving
MeSH Terms: conditions — Cigarette Smoking; Vaping; Smoking

STUDY DESIGN:
Intervention Model Description: All participants will receive all components of this study. Participants receive laboratory sessions in a within-person randomized order. Randomization will determine whether participants receive a cigarette OR e-cigarette cue during the in-vivo cue reactivity task. Participants who receive a given cue during the first laboratory session will receive the other cue during the second session. Within each laboratory session, the presentation order of the trials within the computerized visual dot probe task will also be randomized such that participants will either receive the cigarette vs. neutral OR e-cigarette vs. neutral block first (all participants receive both blocks of trials in both sessions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Protocol (Experimental): All participants will receive all laboratory protocol components in a within-person randomized order across two sequential laboratory sessions.
  Interventions: Behavioral: Cue Reactivity Task; Behavioral: Computerized Visual Dot Probe; Behavioral: Choice Task

INTERVENTIONS:
Behavioral: Cue Reactivity Task — In the cue-reactivity task, participants will be exposed to either a combustible cigarette or e-cigarette cue (within-subjects randomized order across laboratory sessions) and a neutral water bottle cue. Participants will report their craving for cigarettes and e-cigarettes.
Behavioral: Computerized Visual Dot Probe — In the computerized visual dot probe task, participants will view a series of substance (cigarette or e-cigarette by trial block) versus neutral (water bottle) image trials and then respond to a subsequent image presented behind either the neutral or substance image. Order of block presentation within the task is randomized within-subjects across study sessions (i.e., cigarette OR e-cigarette block first).
Behavioral: Choice Task — In the choice task, participants will choose between smoking their usual brand cigarette or their own e-cigarette over ten sequential ad-libbed trials.

SUMMARY:
This study investigates the degree to which shared behavioral processes underlie combustible cigarette (CC) and electronic nicotine delivery system (ENDS) use in young adult dual users of these products in both the laboratory and natural environment. The primary processes examined by this study are cue-reactivity, attentional bias, and affect.

Laboratory hypotheses are: (1) cue exposure will elicit craving of both CC and ENDS in the laboratory and that product-specific cues will elicit stronger craving for the affiliated products; (2) visual probe effects indicating attentional bias in the laboratory will be observed for smoking and vaping images; and (3) cross-conditioning from the first hypothesis will be associated with heaviness of use of CC and ENDS and product choice. Natural environment hypotheses are: (1) presence of tobacco-related cues in the natural environment will elicit craving and use of these products; (2) reactivity to cues, attentional bias, and cross-product conditioning assessed in the laboratory will be associated with craving and use of tobacco products over and above the effects of cues in the natural environment; and (3) negative affect will strengthen these associations.

DETAILED DESCRIPTION:
This project will enroll 80 young adults who regularly use both CC and ENDS. At the start of the study, participants will provide informed consent; biological indicators and self-report measures will be collected; and participants will become enrolled in the study. Participants will then complete two laboratory sessions in a randomized order where they will be: a) exposed to either CC or ENDS cues (based on randomized order) and report their craving for these products; b) complete a computerized attentional bias assessment; and c) choose between smoking their usual brand CC or vaping their own ENDS device over ten sequential opportunities. After the conclusion of the second laboratory session, participants will install a smartphone application that will ask participants questions 5 times per day for 28 days at random intervals assessing: craving for CC and ENDS, physical and social context, affect, and attentional bias. Using the smartphone application, participants will also: a) complete a daily computerized assessment of attentional bias abbreviated from the laboratory sessions; b) report on CC and ENDS cues they experience in the natural environment; and c) report their use of CC and ENDS. A subset of participants will complete a focus group where they will be asked about real-time interventions for smoking and vaping.

Examining these processes in the laboratory and the real world will facilitate: a) evaluating whether behavioral processes related to use and craving in controlled settings operate in similar fashion in naturalistic settings; and b) identifying the situational factors that predict or moderate these effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 34 (inclusive)
* English-speaking at an 8th grade level
* Any self-reported past 7-day use of both ENDS and cigarettes
* Self-identification as a regular ENDS and combustible cigarette user OR use of cigarettes and e-cigarettes on at least 6 of the past 7 days including at least 3 days of using each product;
* Smoking status confirmed via breath CO >= 6 ppm112 or NicAlert test of urine cotinine (level >= 3)
* Smartphone ownership.

Exclusion Criteria:

* Intention to quit smoking or vaping during the next 30 days
* Intention to travel during next 30 days
* Current alcohol dependence (based on MINI)
* Urine-screened or past month illicit substance use other than marijuana (amphetamine, cocaine, methamphetamine, opioids, benzodiazepines
* Pregnant (due to toxicity of tobacco products)
* Current psychosis, mania, or suicidal ideation (based on MINI).

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change in acute craving for cigarettes before and after cue exposure (Session 1) | Laboratory session 1, approximately 1 week after baseline
  Visual analog scale ranging from 0-100. Higher scores = more craving.
Change in acute craving for cigarettes before and after cue exposure (Session 2) | Laboratory session 2, approximately 2 weeks after baseline
  Visual analog scale ranging from 0-100. Higher scores = more craving.
Change in acute craving for e-cigarettes before and after cue exposure (Session 1) | Laboratory session 1, approximately 1 week after baseline
  Visual analog scale ranging from 0-100. Higher scores = more craving.
Change in acute craving for e-cigarettes before and after cue exposure (Session 2) | Laboratory session 2, approximately 2 weeks after baseline
  Visual analog scale ranging from 0-100. Higher scores = more craving.
Change in acute craving for bottled water before and after cue exposure (Session 1) | Laboratory session 1, approximately 1 weeks after baseline
  Visual analog scale ranging from 0-100. Higher scores = more craving.
Change in acute craving for bottled water before and after cue exposure (Session 2) | Laboratory session 2, approximately 2 weeks after baseline
  Visual analog scale ranging from 0-100. Higher scores = more craving.
Attentional bias (objective) (Session 1) | Laboratory session 1, approximately 1 week after baseline
  Mean difference between reaction time of correct responses to visual stimuli presented behind substance-related versus neutral cue. Computed for both cigarettes and e-cigarettes.
Attentional bias (objective) (Session 2) | Laboratory session 2, approximately 2 weeks after baseline
  Mean difference between reaction time of correct responses to visual stimuli presented behind substance-related versus neutral cue. Computed for both cigarettes and e-cigarettes.
Tobacco use (choice) (Session 1) | Laboratory session 1, approximately 1 week after baseline
  Categorical choice between taking a puff of usual brand cigarette, puff from personal ENDS device, or abstaining from either cigarette or ENDS device over ten trials in ad-libbed session lasting 30 minutes. Indexed as any use of product, proportion of trials where product is use, difference between number of trials where each product was used.
Tobacco use (choice) (Session 2) | Laboratory session 2, approximately 2 weeks after baseline
  Categorical choice between taking a puff of usual brand cigarette, puff from personal ENDS device, or abstaining from either cigarette or ENDS device over ten trials in ad-libbed session lasting 30 minutes. Indexed as any use of product, proportion of trials where product is use, difference between number of trials where each product was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data except for transcriptions of focus groups will be made available after the completion of all study activities.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After closing the study IRB protocol and destroying all identifiers. Anticipated 2 years after completion of primary data collection. Data availability will be perpetual. Additional data dissemination plans are pending.